CLINICAL TRIAL: NCT03100747
Title: Evaluating the Role of Incision Height in Trichiasis Surgery Outcomes
Brief Title: Maximizing Trichiasis Surgery Success
Acronym: MTSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Orbis (Other); National Eye Institute (NEI) (NIH); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-2878; UG1EY025992 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-04-04 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Trichiasis; Surgery
MeSH Terms: conditions — Trichiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bilamellar 3 mm (Active Comparator): Bilamellar tarsal rotation trichiasis surgery involves a full-thickness incision through the upper eyelid. For this arm, the height of the incision will be assigned at 3 mm from the eyelid margin.
  Interventions: Procedure: Bilamellar 3 mm
- Bilamellar 5mm (Active Comparator): Bilamellar tarsal rotation trichiasis surgery involves a full-thickness incision through the upper eyelid. For this arm, the height of the incision will be assigned at 5 mm from the eyelid margin.
  Interventions: Procedure: Bilamellar 5 mm
- Trabut 3mm (Active Comparator): Trabut surgery involves a partial-thickness incision through the upper eyelid parallel to the eyelid margin. For this surgery, the height of the incision will be assigned at 3 mm from the eyelid margin.
  Interventions: Procedure: Trabut 3 mm

INTERVENTIONS:
Procedure: Bilamellar 3 mm — Trichiasis surgery using the bilamellar tarsal rotation procedure with incision 3 mm from the eyelid margin
  Other Names: Bilamellar Tarsal Rotation with 3 mm incision
  Arms: Bilamellar 3 mm
Procedure: Bilamellar 5 mm — Trichiasis surgery using the bilamellar tarsal rotation procedure with incision 5 mm from the eyelid margin
  Other Names: Bilamellar Tarsal Rotation with 5mm incision
  Arms: Bilamellar 5mm
Procedure: Trabut 3 mm — Trichiasis surgery using Trabut procedure with incision 3 mm from the eyelid margin
  Other Names: Trabut procedure with 3 mm incision
  Arms: Trabut 3mm

SUMMARY:
The purpose of this study is to determine whether the rate of post-operative trachomatous trichiasis differs significantly between bilamellar tarsal rotation surgery with an incision height of 3 mm, bilamellar tarsal rotation surgery with an incision height of 5 mm, and Trabut surgery.

DETAILED DESCRIPTION:
In this trial the investigators will randomize 4,953 individuals with previously unoperated trichiasis on a 1:1:1 basis to bilamellar tarsal rotation trichiasis surgery with an incision height of 3 mm, bilamellar tarsal rotation trichiasis surgery with an incision height of 5 mm, or Trabut surgery. Participants will receive trichiasis surgery then will be followed at 1 day, 2 weeks, 6 weeks, and 12 months after surgery. Some participants may be asked to attend a follow-up visit at 3-6 months. The primary outcome is development of post-operative trachomatous trichiasis (PTT) within 12 months after surgery. Logistic regression analyses will be performed to compare the rates of PTT in the 3 versus 5 mm incision bilamellar tarsal rotation (BLTR) groups, in the 3 mm BLTR versus Trabut group, and in the 5 mm BLTR versus Trabut group, adjusting for demographic characteristics and pre-operative trichiasis severity.

ELIGIBILITY:
Inclusion Criteria:

* At least one eyelid with previously unoperated upper eyelid trichiasis
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Inability to provide independent, informed consent
* All eyes with previously unoperated trichiasis are phthisical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4914 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Gower, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Orbis Ethiopia, Hosa’ina, Southerns Nations, Nationalities, and Peoples' Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with researchers on an as requested basis after the primary results paper has been published. Interested researchers can contact the principal investigator by email in order to request data and provide a data analysis plan.
Time Frame: 9 to 36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Gower EW, Sisay A, Bayissasse B, Seyum D, Weaver J, Munoz B, Keil AP, Bankoski A, Sullivan KM, Kana H, Admassu F, Tadesse D, Merbs SL. The impact of modified incision height and surgical procedure on trichiasis surgery outcomes: Results of the maximizing trichiasis surgery success (MTSS) randomized trial. PLoS Negl Trop Dis. 2024 Sep 3;18(9):e0012034. doi: 10.1371/journal.pntd.0012034. eCollection 2024 Sep. PMID 39226693
- [Derived] Diallo AO, Bayissasse B, Sisay A, Seyum D, Weaver J, Munoz B, Merbs SL, Gower EW. Effectiveness of Trachomatous Trichiasis Case-identification Approaches in Ethiopia. Epidemiology. 2023 Nov 1;34(6):909-920. doi: 10.1097/EDE.0000000000001656. Epub 2023 Sep 26. PMID 37757880
- [Derived] Bayissasse B, Sullivan KM, Merbs SL, Munoz B, Keil A, Sisay A, Singer A, Gower EW. Maximising trichiasis surgery success (MTSS) trial: rationale and design of a randomised controlled trial to improve trachomatous trichiasis surgical outcomes. BMJ Open. 2020 Mar 18;10(3):e036327. doi: 10.1136/bmjopen-2019-036327. PMID 32193277

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Started | 1631; 2299 eyes | 1648; 2337 eyes | 1635; 2304 eyes
Completed Week 6 | 1514; 2132 eyes | 1498; 2136 eyes | 1518; 2148 eyes
Completed Month 12 | 1467; 2052 eyes | 1478; 2097 eyes | 1468; 2081 eyes
Completed Week 6 and/or Month 12 (End of data collection for the primary outcome.) | 1600; 2257 eyes | 1609; 2290 eyes | 1610; 2268 eyes
Completed Year 3 | 1253; 1760 eyes | 1238; 1757 eyes | 1261; 1781 eyes
Completed | 1253; 1760 eyes | 1238; 1757 eyes | 1261; 1781 eyes
Not Completed | 378; 539 eyes | 410; 580 eyes | 374; 523 eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm | Total
Number analyzed (Participants) | 1631 | 1648 | 1635 | 4914
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 291 | 314 | 311 | 916
  40-60 years | 1075 | 1041 | 1053 | 3169
  > 60 years | 265 | 293 | 271 | 829
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1222 | 1261 | 1223 | 3706
  Male | 409 | 387 | 412 | 1208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1631 | 1648 | 1635 | 4914
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1631 | 1648 | 1635 | 4914
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ethiopia | 1631 | 1648 | 1635 | 4914

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Presence of Post-Operative Trichiasis Within 12 Months
Description: Presence of post-operative trichiasis is defined as 1+ trichiatic eyelashes or evidence of recent epilation. Any eyelashes touching the eye with the eye in primary gaze are considered to be trichiatic. Outcomes will be evaluated at 6 weeks and 12 months. The first date of post-operative trichiasis will be used as the outcome.
Time Frame: 12 Months
Population: Data reported for those participants who completed the Week 6 and/or Month 12 assessment.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1600 | 1609 | 1610
Number analyzed (eyes) | 2257 | 2290 | 2268
eyes | 347 | 504 | 298
Statistical Analysis 1: Comparison: Bilamellar 3 mm vs Trabut 3mm; Test type: Superiority; p = 0.039, Regression, Logistic — The a priori threshold for statistical significance (adjusted for multiple comparisons) is 0.0167; Odds Ratio (OR) = 1.21, 98.3% CI 2-sided [0.97 to 1.52]
Statistical Analysis 2: Comparison: Bilamellar 5mm vs Trabut 3mm; Test type: Superiority; p < 0.0001, Regression, Logistic — The a priori threshold for statistical significance (adjusted for multiple comparisons) is 0.0167; Odds Ratio (OR) = 1.91, 98.3% CI 2-sided [1.54 to 2.36]
Statistical Analysis 3: Comparison: Bilamellar 3 mm vs Bilamellar 5mm; Test type: Superiority; p < 0.0001, Regression, Logistic — The a priori threshold for statistical significance (adjusted for multiple comparisons) is 0.0167; Odds Ratio (OR) = 1.57, 98.3% CI 2-sided [1.29 to 1.92]

2. Secondary Outcome: Number of Eyes With Presence of Post-Operative Trichiasis at 6 Weeks
Description: Presence of post-operative trichiasis is defined as 1+ trichiatic eyelashes or evidence of recent epilation. Any eyelashes touching the eye with the eye in primary gaze are considered to be trichiatic.
Time Frame: 6 Weeks
Population: Data reported only for those participants who completed the Week 6 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1514 | 1498 | 1518
Number analyzed (Eyes) | 2132 | 2136 | 2148
Eyes | 47 | 101 | 59

3. Secondary Outcome: Severity of Post-Operative Trichiasis at 6 Weeks
Description: Severity of post-operative trichiasis will be graded as mild, moderate, or severe based on number of eyelashes touching globe and number of eyelashes epilated.
  Definitions for trichiasis severity are: Mild: 1-4 Eyelashes touching globe, no epilation OR 1-10 Eyelashes epilated, no eyelashes touching globe; Moderate: 5-9 Eyelashes touching globe, no epilation OR 1-4 Eyelashes touching globe and 1-10 eyelashes epilated; Severe: 5-9 Eyelashes touching globe and 1-10 eyelashes epilated OR 10+ Eyelashes touching globe, regardless of epilation status OR 11-20 Eyelashes epilated, regardless of eyelashes touching globe OR Entire eyelid epilated
Time Frame: 6 Weeks
Population: Data reported only for those participants who completed the Week 6 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1514 | 1498 | 1518
Number analyzed (Eyes) | 2132 | 2136 | 2148
Eyes
  None | 2085 | 2035 | 2089
  Mild | 35 | 79 | 42
  Moderate | 8 | 12 | 11
  Severe | 4 | 10 | 6

4. Secondary Outcome: Severity of Post-Operative Trichiasis at 12 Months
Description: as for outcome 3
Time Frame: 12 Months
Population: Data reported only for those participants who completed the Month 12 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1467 | 1478 | 1468
Number analyzed (Eyes) | 2052 | 2097 | 2081
Eyes
  None | 1714 | 1620 | 1801
  Mild | 267 | 348 | 202
  Moderate | 34 | 68 | 44
  Severe | 37 | 61 | 34

5. Secondary Outcome: Number of Eyes With Presence of Eyelid Contour Abnormalities at 6 Weeks
Description: A field and photograph examiner will grade the presence of abnormality independently, using a standardized definition. For this analysis, mild will be combined with normal to create "no significant abnormality" and moderate and severe will be combined into a "moderate/severe contour abnormality" group. The photographic grade will serve as the primary grade for this measure.
  Definitions for abnormality are: Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length; Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length; Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid length
Time Frame: 6 Weeks
Population: Data reported only for those participants who completed the Week 6 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1514 | 1498 | 1518
Number analyzed (Eyes) | 2132 | 2136 | 2148
Eyes
  no significant abnormality | 1748 | 1845 | 1716
  Moderate/severe contour abnormality | 384 | 291 | 432

6. Secondary Outcome: Number of Eyes With Presence of Eyelid Contour Abnormalities Within 12 Months
Description: A field and photograph examiner will grade the presence of abnormality independently. For this analysis, mild is combined with normal to create "no significant abnormality" and moderate and severe are combined into a "moderate/severe contour abnormality" group. The photographic grade will serve as the primary grade. The 12 month dichotomous photograph grade will be the main eyelid contour abnormality (ECA) outcome. Data from the last completed visit (6 weeks or 12 months) are used.
  Definitions for abnormality are: Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length; Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length; Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid length
Time Frame: 12 Months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1600 | 1609 | 1610
Number analyzed (eyes) | 2257 | 2290 | 2268
eyes
  no significant abnormality | 2040 | 2151 | 2015
  moderate/severe contour abnormality | 217 | 139 | 253
Statistical Analysis 1: Comparison: Bilamellar 3 mm vs Trabut 3mm; Test type: Superiority; p = 0.094, Regression, Logistic — p-values adjusted for multiple comparisons; Odds Ratio (OR) = 0.84, 98.3% CI 2-sided [0.65 to 1.08]
Statistical Analysis 2: Comparison: Bilamellar 5mm vs Trabut 3mm; Test type: Superiority; p < 0.0001, Regression, Logistic — p-value adjusted for multiple comparisons, the a priori threshold for statistical significance (adjusted for multiple comparisons) is 0.0167; Odds Ratio (OR) = 0.50, 98.3% CI 2-sided [0.38 to 0.67]
Statistical Analysis 3: Comparison: Bilamellar 3 mm vs Bilamellar 5mm; Test type: Superiority; p < 0.0001, Regression, Logistic — The a priori threshold for statistical significance (adjusted for multiple comparisons) is 0.0167; Odds Ratio (OR) = 0.60, 98.3% CI 2-sided [0.45 to 0.80]

7. Secondary Outcome: Severity of Eyelid Contour Abnormalities at 6 Weeks
Description: Using the grades obtained in the outcome above, the eyelid contour abnormality will be reported as none, mild, moderate, or severe. This is a secondary outcome and will only utilize the photograph grade for this outcome.
  Definitions for abnormality are: Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length; Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length; Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid length
Time Frame: 6 Weeks
Population: Data reported only for those participants who completed the Week 6 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1514 | 1498 | 1518
Number analyzed (Eyes) | 2132 | 2136 | 2148
Eyes
  None | 1465 | 1652 | 1361
  Mild | 283 | 193 | 354
  Moderate | 197 | 127 | 323
  Severe | 187 | 164 | 110

8. Secondary Outcome: Severity of Eyelid Contour Abnormalities at 12 Months
Description: The eyelid contour abnormality will be reported as none, mild, moderate, or severe. This is a secondary outcome and will only utilize the photograph grade for this outcome.
  Definitions for abnormality are: Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length; Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length; Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid length.
Time Frame: 12 Months
Population: Data reported only for those participants who completed the Month 12 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1467 | 1478 | 1468
Number analyzed (Eyes) | 2052 | 2097 | 2081
Eyes
  None | 1780 | 1909 | 1678
  Mild | 90 | 76 | 194
  Moderate | 132 | 79 | 186
  Severe | 50 | 33 | 23

9. Secondary Outcome: Number of Eyes With Changes in Eyelid Contour Abnormalities Between 6 Weeks and 1 Year
Description: The severity of eyelid contour abnormality can lessen over time. The severity will be compared at 6 weeks and 12 months.
Time Frame: 12 months
Population: Only includes participants seen at both 6 weeks and 12 months.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1378 | 1362 | 1374
Number analyzed (Eyes) | 1920 | 1939 | 1956
Eyes
  Better | 183 | 159 | 208
  Same | 1721 | 1769 | 1731
  Worse | 16 | 11 | 17

10. Secondary Outcome: Number of Eyes With Presence of Pyogenic Granuloma at 6 Weeks
Description: Pyogenic granulomas occasionally develop after trichiasis surgery, and it is thought that these are a response to a foreign body, such as suture material or a jagged incision edge. The patient examiners will evaluate presence of granulomas, and all granulomas will be noted, regardless of size.
Time Frame: 6 weeks
Population: Data reported only for those participants who completed the Week 6 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1514 | 1498 | 1518
Number analyzed (Eyes) | 2132 | 2136 | 2148
Eyes | 142 | 109 | 166

11. Secondary Outcome: Number of Eyes With Presence of Pyogenic Granulomas Within 12 Months
Description: Pyogenic granulomas occasionally develop after trichiasis surgery, and it is thought that these are a response to a foreign body, such as suture material or a jagged incision edge. The patient examiners will evaluate presence of granulomas, and all granulomas will be noted, regardless of size. Data are included for both 6 weeks and 12 months.
Time Frame: up to 12 Months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1600 | 1609 | 1610
Number analyzed (Eyes) | 2257 | 2290 | 2268
Eyes | 147 | 118 | 170
Statistical Analysis 1: Comparison: Bilamellar 3 mm vs Trabut 3mm; Test type: Superiority; p = 0.24, Regression, Logistic; Odds Ratio (OR) = 0.86, 98.3% CI 2-sided [0.64 to 1.17]
Statistical Analysis 2: Comparison: Bilamellar 5mm vs Trabut 3mm; Test type: Superiority; p = 0.0037, Regression, Logistic; Odds Ratio (OR) = 0.68, 98.3% CI 2-sided [0.49 to 0.93]
Statistical Analysis 3: Comparison: Bilamellar 3 mm vs Bilamellar 5mm; Test type: Superiority; p = 0.08, Regression, Logistic; Odds Ratio (OR) = 0.78, 98.3% CI 2-sided [0.57 to 1.09]

12. Secondary Outcome: Number of Eyes With Presence of Post-Operative Trichiasis Within 3 Years
Description: Presence of post-operative trichiasis is defined as 1+ trichiatic eyelashes or evidence of recent epilation. Any eyelashes touching the eye with the eye in primary gaze are considered to be trichiatic. Outcomes will be evaluated based on visits at 6 weeks, 12 months and/or Year 3.
Time Frame: up to 3 Years
Population: Data reported for those participants who completed the Week 6, Month 12 and/or Year 3 assessment.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
Number analyzed (Participants) | 1612 | 1622 | 1624
Number analyzed (Eyes) | 2272 | 2305 | 2288
Eyes | 451 | 663 | 401

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 3 year follow-up.
Arm/Group | Bilamellar 3 mm | Bilamellar 5mm | Trabut 3mm
All-Cause Mortality (participants affected / at risk) | 113/1631 | 103/1648 | 102/1635
Serious Adverse Events (participants affected / at risk) | 0/1631 | 1/1648 | 1/1635
Other Adverse Events (participants affected / at risk) | 0/1631 | 0/1648 | 0/1635
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilamellar 3 mm (N=1631) | Bilamellar 5mm (N=1648) | Trabut 3mm (N=1635)
Kidney Stones (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Hospitalization was required due to kidney stones
Whole Body Edema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Whole body edema requiring hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT03100747/Prot_SAP_000.pdf